CLINICAL TRIAL: NCT04673851
Title: Horyzons: Implementation in Clinical Practice
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of North Carolina, Chapel Hill (Other)
Collaborators: North Carolina Department of Health and Human Services (Other Government)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 19-1709
Record Dates: First submitted 2020-12-11; First posted 2020-12-17 (Actual); Results first posted 2024-08-15 (Actual); Last update posted 2024-08-15 (Actual); Status verified 2024-06

CONDITIONS: Schizophrenia; Schizoaffective Disorder; Schizophreniform Disorders; Unspecified Schizophrenia Spectrum and Other Psychotic Disorder
Keywords: Social Media; Virtual Therapeutic Content; First Episode Psychosis; Virtual Therapy
MeSH Terms: conditions — Schizophrenia; Psychotic Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (2):
- FEP Clients (Experimental): Participants with first episode psychosis (FEP) recruited from First Episode Clinics in North Carolina (OASIS, Encompass, Eagle, and SHORE) or UNC-affiliated STEP Clinics (Carr Mill Mall, Vilcom Center, Main Wake Clinic) will participate in the online platform Horyzons for 3 months (cohort 1) or 6 months (cohort 2) as a part of their care plan. Participants will be encouraged to use both the therapeutic content and the moderated online community throughout their time in the study.
  Interventions: Device: Horyzons USA
- FEP Clinicians (Other): Providers (clinicians and peer support specialists) affiliated with First Episode Clinics in North Carolina (OASIS, Encompass, Eagle, and SHORE) will participate in a focus group discussing the implementation and integration of Horyzons into their care routine with clients who participated in the study.
  Interventions: Device: Horyzons USA

INTERVENTIONS:
Device: Horyzons USA — Participants will be oriented to the site (online platform) and how to use it. The site includes curated therapeutic content surrounding issues such as generalized anxiety, social anxiety, social functioning, depression, and distress tolerance. The site also includes a social media function, in which participants and peer support specialists can post text, images, and videos. The site is monitored by graduate students and trained clinicians.

SUMMARY:
A clinical trial investigating the feasibility and acceptability of implementing a moderated online social media platform with therapeutic content, Horyzons, as a part of care received at first-episode psychosis (FEP) clinics across North Carolina. Clients between the ages of 16 and 35 who are enrolled at one of the 4 FEP clinics or 3 UNC-affiliated STEP Clinics in North Carolina will be considered for enrollment in the trial. Cohort 1 participants will have access to the platform for 3 months and cohort 2 participants will have access to the platform for 6 months. All interventions and assessments will be completed virtually/remotely due to the global pandemic.

DETAILED DESCRIPTION:
Purpose: Our primary objective is to examine the feasibility and acceptability of implementing Horyzons as a part of care received at first-episode psychosis clinics across North Carolina. Our primary aim is to understand how to implement a novel treatment approach as part of routine clinical practice with guidance, assistance, and feedback from service providers (e.g., clinicians, peer support specialists) embedded within the clinic. Our second aim is to assess the extent to which clients engage with the platform (i.e., site usage information) and their thoughts and opinions of Horyzons (i.e., feedback and suggestions). Our third aim is to assess change in psychological measures across the three-month (cohort 1) or six-month (cohort 2) study period.

Participants:

Cohort 1:

30 individuals with first episode psychosis (FEP) 20 clinicians and/or peer support specialists from the FEP clinics

Cohort 2:

60 individuals with FEP 20 clinicians and/or peer support specialists from the FEP clinics

Procedures (methods): FEP participants will be recruited over a 16-week period at their respective first episode clinic. Site usage information as well as feedback about their experience will be collected from participants through the Horyzons platform. Site usage information (e.g., number of posts/comments made on the site, the number and types of 'Journeys' or 'Tracks' (therapeutic content) completed by participants, etc.) will be collected automatically through the Horyzons platform. This trial will last three months for cohort 1 and six months for cohort 2. Before being given access to Horyzons, a research assistant, peer support specialist, or clinician will provide instructions and guidance for using the site (i.e., Horyzons induction). Feedback will be collected from participants at the end of the active study period.

Service providers (i.e., clinicians and/or peer support specialists) will be asked to provide feedback about their perceptions of their clients' responses to engaging in Horyzons for the 3-month (cohort 1) or the 6-month (cohort 2) period. Clinicians and peer support specialists will also be asked about their experience integrating the psychosocial intervention in the clinic. Items will include challenges to clinic-wide implementation as well as their feedback to overcome/reduce the impact of these barriers if Horyzons were to be provided as part of routine clinical care in the future. Clinicians and peer support specialists will be interviewed in 1-2 focus groups (depending on schedule and availability) for which these individuals will be compensated.

As Horyzons involves therapeutic content and is designed to improve psychological outcomes such as loneliness and social support, this service is considered part of the clinical care provided to individuals by their respective FEP clinic. As such, participants will not be compensated for their involvement in the platform. Site usage information will be collected automatically through the Horyzons site. However, clients will be compensated for providing feedback about their experience with Horyzons as well as for completing the assessment portion of the study onboarding process.

Finally, Horyzons will be monitored daily (two hours per weekday and one hour per weekend day) by trained peer support specialists, master's level clinicians, and/or graduate students in the Department of Psychology and Neuroscience at UNC. The principal investigator, David Penn, will lead weekly supervision calls to ensure appropriate care and support of clients involved in this project, to discuss case conceptualization and suggestions for engaging clients in the platform, as well as to monitor any potential safety concerns. All clinically-relevant information will be shared with the first episode clinicians involved in participants' mental health care.

ELIGIBILITY:
Inclusion Criteria:

* Clients must be between the ages of 16 and 35
* Clients must have a diagnosis of schizophrenia, schizoaffective disorder, schizophreniform disorder, or Unspecified Schizophrenia Spectrum or Other Psychotic disorder
* Clients must be receiving services at one of the four FEP clinics in North Carolina (OASIS, Encompass, Eagle, or SHORE) or UNC-affiliated STEP clinics (Carr Mill Mall, Vilcom Center, Main Wake Clinic)
* Clients must not have had thoughts of harming themselves in the month before enrollment
* Clients must not have been hospitalized for psychiatric reasons in the three months before enrollment
* Clients must not have had a psychiatric medication change in the month before enrollment
* Clients must have access to the internet through a phone, tablet, or computer

Exclusion Criteria:

* Clients who do not speak English will not be considered for enrollment
* Adult clients (18+ years) with legal guardians (LARs) will not be considered for the study

Ages: 16 Years to 35 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 85 (Actual)
Dates: Start 2021-01-19 (Actual); Primary Completion 2023-08-31 (Actual); Study Completion 2023-08-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David Penn, PhD, Principal Investigator — University of North Carolina, Chapel Hill; Diana Perkins, MD, MPH, Principal Investigator — University of North Carolina, Chapel Hill - School of Medicine
Locations (1):
- University of North Carolina at Chapel Hill, Chapel Hill, North Carolina, United States

IPD SHARING:
Plan to Share IPD: Yes
Deidentified individual data that supports the results will be shared beginning 9 to 36 months following publication provided the investigator who proposes to use the data has approval from an Institutional Review Board (IRB), Independent Ethics Committee (IEC), or Research Ethics Board (REB), as applicable, and executes a data use/sharing agreement with UNC.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: 9 to 36 months following publication
Access Criteria: Requesting investigator has appropriate approval (see above) and an executed data use/sharing agreement with UNC.

REFERENCES:
- [Derived] Pokowitz EL, Stiles BJ, Thomas R, Bullard K, Ludwig KA, Gleeson JF, Alvarez-Jimenez M, Perkins DO, Penn DL. User experiences of an American-adapted moderated online social media platform for first-episode psychosis: Qualitative analysis. Digit Health. 2023 May 22;9:20552076231176700. doi: 10.1177/20552076231176700. eCollection 2023 Jan-Dec. PMID 37252256

RESULTS

PARTICIPANT FLOW:
Groups:
- FEP Clients (Cohort 1): Participants with first episode psychosis (FEP) recruited from First Episode Clinics in North Carolina (OASIS, Encompass, Eagle, and SHORE). Participants will use the online platform Horyzons for 3 months. Participants will be encouraged to use both the therapeutic content and the moderated online community throughout their time in the study.
  Horyzons USA: Participants will be oriented to the site (online platform) and how to use it. The site includes curated therapeutic content surrounding issues such as generalized anxiety, social anxiety, social functioning, depression, and distress tolerance. The site also includes a social media function, in which participants and peer support specialists can post text, images, and videos. The site is monitored by graduate students and trained clinicians.
- FEP Clients (Cohort 2): Participants with first episode psychosis (FEP) recruited from First Episode Clinics in North Carolina (OASIS, Encompass, Eagle, and SHORE). Participants will use the online platform Horyzons for 6 months. Participants will be encouraged to use both the therapeutic content and the moderated online community throughout their time in the study.
  Horyzons USA: Participants will be oriented to the site (online platform) and how to use it. The site includes curated therapeutic content surrounding issues such as generalized anxiety, social anxiety, social functioning, depression, and distress tolerance. The site also includes a social media function, in which participants and peer support specialists can post text, images, and videos. The site is monitored by graduate students and trained clinicians.
- FEP Clinicians (Cohort 1); FEP Clinicians (Cohort 2): Providers (clinicians and peer support specialists) affiliated with First Episode Clinics in North Carolina (OASIS, Encompass, Eagle, and SHORE) will participate in a focus group discussing the implementation and integration of Horyzons into their care routine with clients who participated in the study.
  Horyzons USA: Participants will be oriented to the site (online platform) and how to use it. The site includes curated therapeutic content surrounding issues such as generalized anxiety, social anxiety, social functioning, depression, and distress tolerance. The site also includes a social media function, in which participants and peer support specialists can post text, images, and videos. The site is monitored by graduate students and trained clinicians.
Period: Overall Study
Arm/Group | FEP Clients (Cohort 1) | FEP Clients (Cohort 2) | FEP Clinicians (Cohort 1) | FEP Clinicians (Cohort 2)
Started | 25 | 37 | 12 | 11
Completed | 20 | 27 | 12 | 11
Not Completed | 5 | 10 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- FEP Clients (Cohort 1): Participants with first episode psychosis (FEP) recruited from First Episode Clinics in North Carolina (OASIS, Encompass, Eagle, and SHORE). Participants will use the online platform Horyzons for 3 months as a part of their care plan. Participants will be encouraged to use both the therapeutic content and the moderated online community throughout their time in the study.
  Horyzons USA: Participants will be oriented to the site (online platform) and how to use it. The site includes curated therapeutic content surrounding issues such as generalized anxiety, social anxiety, social functioning, depression, and distress tolerance. The site also includes a social media function, in which participants and peer support specialists can post text, images, and videos. The site is monitored by graduate students and trained clinicians.
- FEP Clients (Cohort 2): Participants with first episode psychosis (FEP) recruited from First Episode Clinics in North Carolina (OASIS, Encompass, Eagle, and SHORE). Participants will use the online platform Horyzons for 6 months as a part of their care plan. Participants will be encouraged to use both the therapeutic content and the moderated online community throughout their time in the study.
  Horyzons USA: Participants will be oriented to the site (online platform) and how to use it. The site includes curated therapeutic content surrounding issues such as generalized anxiety, social anxiety, social functioning, depression, and distress tolerance. The site also includes a social media function, in which participants and peer support specialists can post text, images, and videos. The site is monitored by graduate students and trained clinicians.
- Total: Total of all reporting groups
Arm/Group | FEP Clients (Cohort 1) | FEP Clients (Cohort 2) | FEP Clinicians (Cohort 1) | FEP Clinicians (Cohort 2) | Total
Number analyzed (Participants) | 25 | 37 | 12 | 11 | 85
Age, Continuous [Mean (Standard Deviation); unit: years] — Population: Number analyzed in row differs from overall due to missing data.
  years
    number analyzed (Participants) | 25 | 37 | 12 | 9 | 83
    (all) | 24.88 (4.58) | 22.76 (4.56) | 41.75 (15.00) | 40.67 (15.06) | 28.08 (11.32)
Sex/Gender, Customized [Count of Participants; unit: Participants] — Population: Number analyzed in row differs from overall due to missing data.
  Participants
    Female: number analyzed (Participants) | 25 | 37 | 12 | 10 | 84
    Female | 6 | 12 | 8 | 8 | 34
    Male: number analyzed (Participants) | 25 | 37 | 12 | 10 | 84
    Male | 19 | 24 | 3 | 1 | 47
    Non-Binary: number analyzed (Participants) | 25 | 37 | 12 | 10 | 84
    Non-Binary | 0 | 1 | 1 | 1 | 3
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants] — Population: Number analyzed in row differs from overall due to missing data.
  Participants
    number analyzed (Participants) | 25 | 37 | 12 | 10 | 84
    Hispanic or Latino | 3 | 2 | 0 | 0 | 5
    Not Hispanic or Latino | 22 | 35 | 12 | 9 | 78
    Unknown or Not Reported | 0 | 0 | 0 | 1 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants] — Population: Number analyzed in row differs from overall due to missing data.
  Participants
    number analyzed (Participants) | 25 | 37 | 12 | 10 | 84
    American Indian or Alaska Native | 1 | 1 | 0 | 0 | 2
    Asian | 1 | 3 | 0 | 0 | 4
    Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
    Black or African American | 6 | 11 | 3 | 0 | 20
    White | 16 | 15 | 9 | 9 | 49
    More than one race | 0 | 7 | 0 | 1 | 8
    Unknown or Not Reported | 1 | 0 | 0 | 0 | 1
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 25 | 37 | 12 | 11 | 85
Participant Education Level [Count of Participants; unit: Participants] — Population: Number analyzed in row differs from overall due to missing data.
  Participants
    number analyzed (Participants) | 25 | 37 | 12 | 10 | 84
    Middle school or less | 0 | 0 | 0 | 0 | 0
    Some high school | 2 | 3 | 0 | 0 | 5
    High school diploma or equivalent | 4 | 12 | 0 | 0 | 16
    Some college | 12 | 14 | 1 | 1 | 28
    College degree | 6 | 7 | 1 | 0 | 14
    Higher than college | 1 | 1 | 10 | 9 | 21
Years of Education [Mean (Standard Deviation); unit: years] — Population: Number analyzed in row differs from overall due to missing data.
  years
    number analyzed (Participants) | 25 | 37 | 12 | 5 | 79
    (all) | 14.16 (2.89) | 13.49 (1.86) | 19.75 (2.98) | 20 (2.92) | 15.06 (3.50)
Diagnosis [Count of Participants; unit: Participants] — Population: Data not applicable to FEP Clinicians and therefore not collected for this group.
  Participants
    number analyzed (Participants) | 25 | 37 | 0 | 0 | 62
    Schizophrenia | 9 | 18 |  |  | 27
    Schizoaffective disorder | 7 | 6 |  |  | 13
    Schizophreniform disorder | 1 | 1 |  |  | 2
    Brief psychotic disorder | 0 | 1 |  |  | 1
    Schizotypal personality disorder | 1 | 0 |  |  | 1
    Bipolar disorder with psychotic features | 1 | 4 |  |  | 5
    Major depressive disorder with psychotic features | 0 | 1 |  |  | 1
    Substance-induced psychotic disorder | 1 | 0 |  |  | 1
    Unspecified psychotic disorder | 5 | 6 |  |  | 11
    Unknown/Not Reported | 0 | 0 |  |  | 0
Age at Diagnosis of Psychotic Illness [Mean (Standard Deviation); unit: years] — Population: Data not applicable to FEP Clinicians and therefore not collected for this group. Number analyzed in row differs from overall due to missing data.
  years
    number analyzed (Participants) | 25 | 34 | 0 | 0 | 59
    (all) | 21.24 (3.52) | 19.68 (4.57) |  |  | 20.34 (4.20)
Duration of Psychotic Illness Prior to Study Entry [Mean (Standard Deviation); unit: years] — Population: Data not applicable to FEP Clinicians and therefore not collected for this group. Number analyzed in row differs from overall due to missing data.
  years
    number analyzed (Participants) | 25 | 34 | 0 | 0 | 59
    (all) | 4.20 (2.81) | 3.24 (3.05) |  |  | 3.64 (2.96)
Duration of Untreated Psychotic Illness Prior to Study Entry [Mean (Standard Deviation); unit: years] — Population: Data not applicable to FEP Clinicians and therefore not collected for this group. Number analyzed in row differs from overall due to missing data.
  years
    number analyzed (Participants) | 24 | 34 | 0 | 0 | 58
    (all) | 0.38 (0.66) | 0.49 (0.67) |  |  | 0.45 (0.66)
Number of Lifetime Hospitalizations Prior to Study Entry [Median (Full Range); unit: hospitalizations] — Population: Data not applicable to FEP Clinicians and therefore not collected for this group. Number analyzed in row differs from overall due to missing data.
  hospitalizations
    number analyzed (Participants) | 25 | 36 | 0 | 0 | 61
    (all) | 2 [0 to 5] | 1 [0 to 10] |  |  | 2 [0 to 10]

OUTCOME MEASURES:

1. Primary Outcome: Mean Change in UCLA Loneliness Scale Score (Both Cohorts)
Description: The UCLA Loneliness scale is a 20 item scale. Answers are on a 4 point scale with options "I often feel this way," "I sometimes feel this way," "I rarely feel this way," and "I never feel this way." Possible scores range from 20 to 80. Higher scores reflect worse outcomes (greater feelings of loneliness). The UCLA Loneliness Scale is a part of the PhenX Toolkit. The UCLA Loneliness Scale is administered in both cohort 1 (Baseline, Mid-treatment, Post-treatment, up to 3 months) and cohort 2 (Baseline, Mid-treatment, Post-treatment, up to 6 months).
Time Frame: Cohort 1: Baseline, Mid-treatment (single assessment between Month 1-2), and Post-treatment (up to 3 months); Cohort 2: Baseline, Mid-treatment (single assessment between Month 2-4), and Post-treatment (up to 6 months)
Population: This outcome only applies to FEP Clients. Mid- and post-treatment data were unavailable for participants who withdrew or were lost to follow-up (Mid-treatment: n = 4 in cohort 1, n = 7 in cohort 2; Post-treatment: n = 5 in cohort 1; n = 10 in cohort 2).
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | FEP Clients (Cohort 1) | FEP Clients (Cohort 2)
Number analyzed (Participants) | 25 | 37
score on a scale
  Baseline | 42.96 (11.64) | 45.08 (11.53)
  Mid-treatment: number analyzed (Participants) | 21 | 30
  Mid-treatment | 41.95 (12.84) | 42.47 (10.75)
  Post-treatment: number analyzed (Participants) | 20 | 27
  Post-treatment | 39.70 (13.70) | 40.78 (12.67)
Statistical Analysis 1: Comparison: FEP Clients (Cohort 1); Midtreatment - Baseline: 21 participants analyzed (had data at both timepoints); Test type: Other — Single group mean difference between baseline and mid-treatment assessments; Mean Difference (Net) = -0.86, Standard Deviation 5.44
Statistical Analysis 2: Comparison: FEP Clients (Cohort 1); Midtreatment - Baseline: 21 participants analyzed (had data at both timepoints); Test type: Other — Effect size of single group mean difference between baseline and mid-treatment assessments; Cohen's d = 0.16
Statistical Analysis 3: Comparison: FEP Clients (Cohort 1); Posttreatment - Baseline: 20 participants analyzed (had data at both timepoints); Test type: Other — Single group mean difference between baseline and post-treatment assessments; Mean Difference (Net) = -2.65, Standard Deviation 5.61
Statistical Analysis 4: Comparison: FEP Clients (Cohort 1); Posttreatment - Baseline: 20 participants analyzed (had data at both timepoints); Test type: Other — Effect size of single group mean difference between baseline and post-treatment assessments; Cohen's d = 0.47
Statistical Analysis 5: Comparison: FEP Clients (Cohort 2); Midtreatment - Baseline: 30 participants analyzed (had data at both timepoints); Test type: Other — Single group mean difference between baseline and mid-treatment assessments; Mean Difference (Net) = -1.97, Standard Deviation 7.19
Statistical Analysis 6: Comparison: FEP Clients (Cohort 2); Midtreatment - Baseline: 30 participants analyzed (had data at both timepoints); Test type: Other — Effect size of single group mean difference between baseline and mid-treatment assessments; Cohen's d = 0.27
Statistical Analysis 7: Comparison: FEP Clients (Cohort 2); Posttreatment - Baseline: 27 participants analyzed (had data at both timepoints); Test type: Other — Single group mean difference between baseline and post-treatment assessments; Mean Difference (Net) = -4.15, Standard Deviation 7.93
Statistical Analysis 8: Comparison: FEP Clients (Cohort 2); Posttreatment - Baseline: 27 participants analyzed (had data at both timepoints); Test type: Other — Effect size of single group mean difference between baseline and post-treatment assessments; Cohen's d = 0.52

2. Primary Outcome: Mean Change in Medical Outcomes Study (MOS) Social Support Survey - Total Score (Both Cohorts)
Description: The MOS Social Support Survey is a 19 item scale. Answers are on a 5 point scale with options "none of the time", "a little of the time", "some of the time", "most of the time", and "all of the time". Possible scores range from 19 to 95. Higher scores reflect higher feelings of social support (more perceived social support). The MOS Social Support Survey is a part of the PhenX Toolkit. The MOS Social Support Survey is administered in both cohort 1 (Baseline, Mid-treatment, Post-treatment, up to 3 months) and cohort 2 (Baseline, Mid-treatment, Post-treatment, up to 6 months).
Time Frame: as for outcome 1
Population: This outcome only applies to FEP Clients. Mid- and post-treatment data were not available for participants who withdrew or were lost to follow-up (Mid-treatment: n = 4 in cohort 1, n = 7 in cohort 2; Post-treatment: n = 5 in cohort 1; n = 10 in cohort 2).
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | FEP Clients (Cohort 1) | FEP Clients (Cohort 2)
Number analyzed (Participants) | 25 | 37
score on a scale
  Baseline | 77.28 (12.36) | 73.24 (15.22)
  Mid-treatment: number analyzed (Participants) | 21 | 30
  Mid-treatment | 76.19 (12.29) | 74.90 (14.16)
  Post-treatment: number analyzed (Participants) | 20 | 27
  Post-treatment | 79.45 (9.68) | 76.59 (14.45)
Statistical Analysis 1: Comparison: FEP Clients (Cohort 1); Midtreatment - Baseline: 21 participants analyzed (had data at both timepoints); Test type: Other — Single group mean difference between baseline and mid-treatment assessments; Mean Difference (Net) = -1.52, Standard Deviation 8.95
Statistical Analysis 2: Comparison: FEP Clients (Cohort 1); Midtreatment - Baseline: 21 participants analyzed (had data at both timepoints); Test type: Other — Effect size of single group mean difference between baseline and mid-treatment assessments; Cohen's d = 0.17
Statistical Analysis 3: Comparison: FEP Clients (Cohort 1); Posttreatment - Baseline: 20 participants analyzed (had data at both timepoints); Test type: Other — Single group mean difference between baseline and post-treatment assessments; Mean Difference (Net) = 1.15, Standard Deviation 5.80
Statistical Analysis 4: Comparison: FEP Clients (Cohort 1); Posttreatment - Baseline: 20 participants analyzed (had data at both timepoints); Test type: Other — Effect size of single group mean difference between baseline and post-treatment assessments; Cohen's d = 0.20
Statistical Analysis 5: Comparison: FEP Clients (Cohort 2); Midtreatment - Baseline: 30 participants analyzed (had data at both timepoints); Test type: Other — Single group mean difference between baseline and mid-treatment assessments; Mean Difference (Net) = 0.67, Standard Deviation 10.29
Statistical Analysis 6: Comparison: FEP Clients (Cohort 2); Midtreatment - Baseline: 30 participants analyzed (had data at both timepoints); Test type: Other — Effect size of single group mean difference between baseline and mid-treatment assessments; Cohen's d = 0.07
Statistical Analysis 7: Comparison: FEP Clients (Cohort 2); Posttreatment - Baseline: 27 participants analyzed (had data at both timepoints); Test type: Other — Single group mean difference between baseline and post-treatment assessments; Mean Difference (Net) = 2.07, Standard Deviation 9.47
Statistical Analysis 8: Comparison: FEP Clients (Cohort 2); Posttreatment - Baseline: 27 participants analyzed (had data at both timepoints); Test type: Other — Effect size of single group mean difference between baseline and post-treatment assessments; Cohen's d = 0.22

3. Secondary Outcome: Mean Change in Social Interaction Anxiety Scale (SIAS) Score (Both Cohorts)
Description: The Social Interaction Anxiety Scale (SIAS) is a 20 item scale. Answers are on a 5-point scale starting at 0 with options "none at all", "slightly", "moderately", "very", and "extremely". Possible scores range from 0 to 80. Higher scores reflect higher levels of social anxiety. Scoring a 43 or higher may indicate a diagnosis of social anxiety, and scores between 34 and 42 may indicate social phobia(s). The SIAS is administered in both cohort 1 (Baseline, Mid-treatment, Post-treatment, up to 3 months) and cohort 2 (Baseline, Mid-treatment, Post-treatment, up to 6 months).
Time Frame: as for outcome 1
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | FEP Clients (Cohort 1) | FEP Clients (Cohort 2)
Number analyzed (Participants) | 25 | 37
score on a scale
  Baseline | 26.24 (11.23) | 27.54 (15.97)
  Mid-treatment: number analyzed (Participants) | 21 | 30
  Mid-treatment | 26.90 (13.58) | 28.90 (18.61)
  Post-treatment: number analyzed (Participants) | 20 | 27
  Post-treatment | 23.85 (13.97) | 26.85 (18.65)
Statistical Analysis 1: Comparison: FEP Clients (Cohort 1); Midtreatment - Baseline: 21 participants analyzed (had data at both timepoints); Test type: Other — Single group mean difference between baseline and mid-treatment assessments; Mean Difference (Net) = -0.05, Standard Deviation 7.08
Statistical Analysis 2: Comparison: FEP Clients (Cohort 1); Midtreatment - Baseline: 21 participants analyzed (had data at both timepoints); Test type: Other — Effect size of single group mean difference between baseline and mid-treatment assessments; Cohen's d = 0.01
Statistical Analysis 3: Comparison: FEP Clients (Cohort 1); Posttreatment - Baseline: 20 participants analyzed (had data at both timepoints); Test type: Other — Single group mean difference between baseline and post-treatment assessments; Mean Difference (Net) = -2.35, Standard Deviation 7.53
Statistical Analysis 4: Comparison: FEP Clients (Cohort 1); Posttreatment - Baseline: 20 participants analyzed (had data at both timepoints); Test type: Other — Effect size of single group mean difference between baseline and post-treatment assessments; Cohen's d = 0.31
Statistical Analysis 5: Comparison: FEP Clients (Cohort 2); Midtreatment - Baseline: 30 participants analyzed (had data at both timepoints); Test type: Other — Single group mean difference between baseline and mid-treatment assessments; Mean Difference (Net) = 0.90, Standard Deviation 9.95
Statistical Analysis 6: Comparison: FEP Clients (Cohort 2); Midtreatment - Baseline: 30 participants analyzed (had data at both timepoints); Test type: Other — Effect size of single group mean difference between baseline and mid-treatment assessments; Cohen's d = 0.09
Statistical Analysis 7: Comparison: FEP Clients (Cohort 2); Posttreatment - Baseline: 27 participants analyzed (had data at both timepoints); Test type: Other — Single group mean difference between baseline and post-treatment assessments; Mean Difference (Net) = -2.56, Standard Deviation 9.60
Statistical Analysis 8: Comparison: FEP Clients (Cohort 2); Posttreatment - Baseline: 27 participants analyzed (had data at both timepoints); Test type: Other — Effect size of single group mean difference between baseline and post-treatment assessments; Cohen's d = 0.27

4. Secondary Outcome: Mean Change in Psychological Wellbeing Scale Short Form - Total Score (Both Cohorts)
Description: The Psychological Wellbeing Scale (Short Form) is an 18 item scale. Answers are on a 6 point scale with options "strongly disagree", "moderately disagree", "slightly disagree", "slightly agree", "moderately agree", and "strongly agree". Possible scores range from 18 to 108. Higher scores reflect higher levels of psychological wellbeing. The Psychological Wellbeing Scale is administered in both cohort 1 (Baseline, Mid-treatment, Post-treatment, up to 3 months) and cohort 2 (Baseline, Mid-treatment, Post-treatment, up to 6 months).
Time Frame: as for outcome 1
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | FEP Clients (Cohort 1) | FEP Clients (Cohort 2)
Number analyzed (Participants) | 25 | 37
score on a scale
  Baseline | 83.80 (14.54) | 78.38 (14.80)
  Mid-treatment: number analyzed (Participants) | 21 | 30
  Mid-treatment | 84.57 (14.68) | 81.87 (14.95)
  Post-treatment: number analyzed (Participants) | 20 | 27
  Post-treatment | 88.20 (15.94) | 86.41 (15.33)
Statistical Analysis 1: Comparison: FEP Clients (Cohort 1); Midtreatment - Baseline: 21 participants analyzed (had data at both timepoints); Test type: Other — Single group mean difference between baseline and mid-treatment assessments; Mean Difference (Net) = -0.29, Standard Deviation 8.27
Statistical Analysis 2: Comparison: FEP Clients (Cohort 1); Midtreatment - Baseline: 21 participants analyzed (had data at both timepoints); Test type: Other — Effect size of single group mean difference between baseline and mid-treatment assessments; Cohen's d = 0.04
Statistical Analysis 3: Comparison: FEP Clients (Cohort 1); Posttreatment - Baseline: 20 participants analyzed (had data at both timepoints); Test type: Other — Single group mean difference between baseline and post-treatment assessments; Mean Difference (Net) = 2.60, Standard Deviation 7.86
Statistical Analysis 4: Comparison: FEP Clients (Cohort 1); Posttreatment - Baseline: 20 participants analyzed (had data at both timepoints); Test type: Other — Effect size of single group mean difference between baseline and post-treatment assessments; Cohen's d = 0.33
Statistical Analysis 5: Comparison: FEP Clients (Cohort 2); Midtreatment - Baseline: 30 participants analyzed (had data at both timepoints); Test type: Other — Single group mean difference between baseline and mid-treatment assessments; Mean Difference (Net) = 2.17, Standard Deviation 7.84
Statistical Analysis 6: Comparison: FEP Clients (Cohort 2); Midtreatment - Baseline: 30 participants analyzed (had data at both timepoints); Test type: Other — Effect size of single group mean difference between baseline and mid-treatment assessments; Cohen's d = 0.28
Statistical Analysis 7: Comparison: FEP Clients (Cohort 2); Posttreatment - Baseline: 27 participants analyzed (had data at both timepoints); Test type: Other — Single group mean difference between baseline and post-treatment assessments; Mean Difference (Net) = 6.48, Standard Deviation 8.50
Statistical Analysis 8: Comparison: FEP Clients (Cohort 2); Posttreatment - Baseline: 27 participants analyzed (had data at both timepoints); Test type: Other — Effect size of single group mean difference between baseline and post-treatment assessments; Cohen's d = 0.76

5. Other Pre Specified Outcome: Mean Change in Working Alliance Inventory for Guided Internet Interventions - Total Score (Both Cohorts)
Description: The Working Alliance Inventory for Guided Internet Interventions (WAI-I) - Total Score is a 12-item scale. Answers are on a 5-point scale with options "seldom", "sometimes", "fairly often", "very often", and "always". Possible scores range from 12 to 60 (summed). Higher scores reflect greater therapeutic alliance. The WAI-I is administered in both cohort 1 (Mid-treatment, Post-treatment, up to 3 months) and cohort 2 (1.5 Months, Mid-treatment, 4.5 Months, Post-treatment, up to 6 months).
Time Frame: Cohort 1: Mid-treatment (between Month 1-2), Post-treatment (up to 3 months); Cohort 2: 1.5 months (between Month 1-2), Mid-treatment (between Month 2-4), 4.5 months (between Month 4-5), Post-treatment (up to 6 months)
Population: This outcome only applies to FEP Clients. Data were not available for participants who withdrew or were lost to follow-up (1.5-month assessment [cohort 2 only]: n = 5; Mid-treatment: n = 4 in cohort 1, n = 7 in cohort 2; 4.5-month assessment [cohort 2 only]: n = 10; Post-treatment: n = 5 in cohort 1; n = 10 in cohort 2). As per protocol, the 1.5 and 4.5 month assessments were not performed for Cohort 1.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | FEP Clients (Cohort 1) | FEP Clients (Cohort 2)
Number analyzed (Participants) | 21 | 32
score on a scale
  1.5 months: number analyzed (Participants) | 0 | 32
  1.5 months |  | 49.75 (7.36)
  Mid-treatment: number analyzed (Participants) | 21 | 30
  Mid-treatment | 45.81 (8.26) | 50.33 (9.09)
  4.5 months: number analyzed (Participants) | 0 | 27
  4.5 months |  | 49.15 (7.44)
  Post-treatment: number analyzed (Participants) | 20 | 27
  Post-treatment | 49.80 (7.88) | 46.41 (9.75)
Statistical Analysis 1: Comparison: FEP Clients (Cohort 1); Posttreatment - Midtreatment: 19 participants analyzed (had data at both timepoints); Test type: Other — Single group mean difference between mid-treatment and post-treatment assessments; Mean Difference (Net) = 4.11, Standard Deviation 6.86
Statistical Analysis 2: Comparison: FEP Clients (Cohort 1); Posttreatment - Midtreatment: 19 participants analyzed (had data at both timepoints); Test type: Other — Effect size of single group mean difference between mid-treatment and post-treatment assessments; Cohen's d = 0.60
Statistical Analysis 3: Comparison: FEP Clients (Cohort 2); Midtreatment - 1.5 Months: 30 participants analyzed (had data at both timepoints); Test type: Other — Single group mean difference between 1.5 month and mid-treatment assessments; Mean Difference (Net) = 0.77, Standard Deviation 6.88
Statistical Analysis 4: Comparison: FEP Clients (Cohort 2); Midtreatment - 1.5 Months: 30 participants analyzed (had data at both timepoints); Test type: Other — Effect size of single group mean difference between 1.5 month and mid-treatment assessments; Cohen's d = 0.11
Statistical Analysis 5: Comparison: FEP Clients (Cohort 2); 4.5 Months - 1.5 Months: 27 participants analyzed (had data at both timepoints); Test type: Other — Single group mean difference between 1.5 month and 4.5 month assessments; Mean Difference (Net) = -0.15, Standard Deviation 5.78
Statistical Analysis 6: Comparison: FEP Clients (Cohort 2); 4.5 Months - 1.5 Months: 27 participants analyzed (had data at both timepoints); Test type: Other — Effect size of single group mean difference between 1.5 month and 4.5 month assessments; Cohen's d = 0.03
Statistical Analysis 7: Comparison: FEP Clients (Cohort 2); Posttreatment - 1.5 Months: 27 participants analyzed (had data at both timepoints); Test type: Other — Single group mean difference between 1.5 month and post-treatment assessments; Mean Difference (Net) = -2.63, Standard Deviation 7.95
Statistical Analysis 8: Comparison: FEP Clients (Cohort 2); Posttreatment - 1.5 Months: 27 participants analyzed (had data at both timepoints); Test type: Other — Effect size of single group mean difference between 1.5 month and post-treatment assessments; Cohen's d = 0.33

6. Other Pre Specified Outcome: Mean Change in Working Alliance Inventory for Guided Internet Interventions - Bond Subscale Score (Both Cohorts)
Description: The Working Alliance Inventory for Guided Internet Interventions - Bond subscale score is a 4-item scale. Answers are on a 5-point scale with options "seldom", "sometimes", "fairly often", "very often", and "always". Possible scores range from 4 to 20 (summed). Higher scores reflect greater bond with a clinician. The WAI-I - Bond subscale is administered in both cohort 1 (Mid-treatment, Post-treatment, up to 3 months) and cohort 2 (1.5 Months, Mid-treatment, 4.5 Months, Post-treatment, up to 6 months).
Time Frame: as for outcome 5
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | FEP Clients (Cohort 1) | FEP Clients (Cohort 2)
Number analyzed (Participants) | 21 | 32
score on a scale
  1.5 months: number analyzed (Participants) | 0 | 32
  1.5 months |  | 18.56 (2.05)
  Mid-treatment: number analyzed (Participants) | 21 | 30
  Mid-treatment | 16.86 (4.05) | 18.50 (2.81)
  4.5 months: number analyzed (Participants) | 0 | 27
  4.5 months |  | 18.00 (2.56)
  Post-treatment: number analyzed (Participants) | 20 | 27
  Post-treatment | 18.50 (2.12) | 17.93 (2.63)
Statistical Analysis 1: Comparison: FEP Clients (Cohort 1); Posttreatment - Midtreatment: 19 participants analyzed (had data at both timepoints); Test type: Other — Single group mean difference between mid-treatment and post-treatment assessments; Mean Difference (Net) = 1.68, Standard Deviation 3.76
Statistical Analysis 2: Comparison: FEP Clients (Cohort 1); Posttreatment - Midtreatment: 19 participants analyzed (had data at both timepoints); Test type: Other — Effect size of single group mean difference between mid-treatment and post-treatment assessments; Cohen's d = 0.45
Statistical Analysis 3: Comparison: FEP Clients (Cohort 2); Midtreatment - 1.5 Months: 30 participants analyzed (had data at both timepoints); Test type: Other — Single group mean difference between 1.5 month and mid-treatment assessments; Mean Difference (Net) = -0.07, Standard Deviation 2.73
Statistical Analysis 4: Comparison: FEP Clients (Cohort 2); Midtreatment - 1.5 Months: 30 participants analyzed (had data at both timepoints); Test type: Other — Effect size of single group mean difference between 1.5 month and mid-treatment assessments; Cohen's d = 0.02
Statistical Analysis 5: Comparison: FEP Clients (Cohort 2); 4.5 Months - 1.5 Months: 27 participants analyzed (had data at both timepoints); Test type: Other — Single group mean difference between 1.5 month and 4.5 month assessments; Mean Difference (Net) = -0.56, Standard Deviation 2.44
Statistical Analysis 6: Comparison: FEP Clients (Cohort 2); 4.5 Months - 1.5 Months: 27 participants analyzed (had data at both timepoints); Test type: Other — Effect size of single group mean difference between 1.5 month and 4.5 month assessments; Cohen's d = 0.23
Statistical Analysis 7: Comparison: FEP Clients (Cohort 2); Posttreatment - 1.5 Months: 27 participants analyzed (had data at both timepoints); Test type: Other — Single group mean difference between 1.5 month and post-treatment assessments; Mean Difference (Net) = -0.59, Standard Deviation 3.15
Statistical Analysis 8: Comparison: FEP Clients (Cohort 2); Posttreatment - 1.5 Months: 27 participants analyzed (had data at both timepoints); Test type: Other — Effect size of single group mean difference between 1.5 month and post-treatment assessments; Cohen's d = 0.19

7. Other Pre Specified Outcome: Mean Change in Working Alliance Inventory for Guided Internet Interventions - Goal/Task Subscale Score (Both Cohorts)
Description: The Working Alliance Inventory for Guided Internet Interventions - Goal/Task Score is an 8-item scale. Answers are on a 5-point scale with options "seldom", "sometimes", "fairly often", "very often", and "always". Possible scores range from 8 to 40 (summed). Higher scores reflect greater shared goals and tasks with a clinician. The WAI-I - Goal/Task subscale is administered in both cohort 1 (Mid-treatment, Post-treatment, up to 3 months) and cohort 2 (1.5 Months, Mid-treatment, 4.5 Months, Post-treatment, up to 6 months).
Time Frame: as for outcome 5
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | FEP Clients (Cohort 1) | FEP Clients (Cohort 2)
Number analyzed (Participants) | 21 | 32
score on a scale
  1.5 months: number analyzed (Participants) | 0 | 32
  1.5 months |  | 31.19 (6.03)
  Mid-treatment: number analyzed (Participants) | 21 | 30
  Mid-treatment | 28.95 (5.50) | 31.83 (6.86)
  4.5 months: number analyzed (Participants) | 0 | 27
  4.5 months |  | 31.15 (5.78)
  Post-treatment: number analyzed (Participants) | 20 | 27
  Post-treatment | 31.30 (6.33) | 28.48 (7.93)
Statistical Analysis 1: Comparison: FEP Clients (Cohort 1); Posttreatment - Midtreatment: 19 participants analyzed (had data at both timepoints); Test type: Other — Single group mean difference between mid-treatment and post-treatment assessments; Mean Difference (Net) = 2.42, Standard Deviation 4.48
Statistical Analysis 2: Comparison: FEP Clients (Cohort 1); Posttreatment - Midtreatment: 19 participants analyzed (had data at both timepoints); Test type: Other — Effect size of single group mean difference between mid-treatment and post-treatment assessments; Cohen's d = 0.54
Statistical Analysis 3: Comparison: FEP Clients (Cohort 2); Midtreatment - 1.5 Months: 30 participants analyzed (had data at both timepoints); Test type: Other — Single group mean difference between 1.5 month and mid-treatment assessments; Mean Difference (Net) = 0.83, Standard Deviation 5.05
Statistical Analysis 4: Comparison: FEP Clients (Cohort 2); Midtreatment - 1.5 Months: 30 participants analyzed (had data at both timepoints); Test type: Other — Effect size of single group mean difference between 1.5 month and mid-treatment assessments; Cohen's d = 0.17
Statistical Analysis 5: Comparison: FEP Clients (Cohort 2); 4.5 Months - 1.5 Months: 27 participants analyzed (had data at both timepoints); Test type: Other — Single group mean difference between 1.5 month and 4.5 month assessments; Mean Difference (Net) = 0.41, Standard Deviation 4.55
Statistical Analysis 6: Comparison: FEP Clients (Cohort 2); 4.5 Months - 1.5 Months: 27 participants analyzed (had data at both timepoints); Test type: Other — Effect size of single group mean difference between 1.5 month and 4.5 month assessments; Cohen's d = 0.09
Statistical Analysis 7: Comparison: FEP Clients (Cohort 2); Posttreatment - 1.5 Months: 27 participants analyzed (had data at both timepoints); Test type: Other — Single group mean difference between 1.5 month and post-treatment assessments; Mean Difference (Net) = -2.04, Standard Deviation 6.12
Statistical Analysis 8: Comparison: FEP Clients (Cohort 2); Posttreatment - 1.5 Months: 27 participants analyzed (had data at both timepoints); Test type: Other — Effect size of single group mean difference between 1.5 month and post-treatment assessments; Cohen's d = 0.33

8. Other Pre Specified Outcome: Mean Change in Medical Outcomes Study (MOS) Social Support Survey - Emotional/Informational Support Subscale Score (Both Cohorts)
Description: The MOS Social Support Survey - Emotional/informational support subscale is an 8 item subscale. Answers are on a 5 point scale with options "none of the time", "a little of the time", "some of the time", "most of the time", and "all of the time". Possible scores range from 8 to 40. Higher scores reflect higher feelings of emotional and informational social support (more perceived emotional and informational social support). The MOS Social Support Survey - Emotional/informational support subscale is administered in both cohort 1 (Baseline, Mid-treatment, Post-treatment, up to 3 months) and cohort 2 (Baseline, Mid-treatment, Post-treatment, up to 6 months).
Time Frame: up to 6 months
Reporting Status: Not Posted

9. Other Pre Specified Outcome: Mean Change in Medical Outcomes Study (MOS) Social Support Survey - Tangible Support Subscale Score (Both Cohorts)
Description: The MOS Social Support Survey - Tangible support subscale is a 4 item subscale. Answers are on a 5 point scale with options "none of the time", "a little of the time", "some of the time", "most of the time", and "all of the time". Possible scores range from 4 to 20. Higher scores reflect higher feelings of tangible social support (more perceived tangible social support). The MOS Social Support Survey - Tangible support subscale is administered in both cohort 1 (Baseline, Mid-treatment, Post-treatment, up to 3 months) and cohort 2 (Baseline, Mid-treatment, Post-treatment, up to 6 months).
Time Frame: up to 6 months
Reporting Status: Not Posted

10. Other Pre Specified Outcome: Mean Change in Medical Outcomes Study (MOS) Social Support Survey - Affectionate Support Subscale Score (Both Cohorts)
Description: The MOS Social Support Survey - Affectionate support subscale is a 3 item subscale. Answers are on a 5 point scale with options "none of the time", "a little of the time", "some of the time", "most of the time", and "all of the time". Possible scores range from 3 to 15. Higher scores reflect higher feelings of affectionate social support (more perceived affectionate social support). The MOS Social Support Survey - Affectionate support subscale is administered in both cohort 1 (Baseline, Mid-treatment, Post-treatment, up to 3 months) and cohort 2 (Baseline, Mid-treatment, Post-treatment, up to 6 months).
Time Frame: up to 6 months
Reporting Status: Not Posted

11. Other Pre Specified Outcome: Mean Change in Medical Outcomes Study (MOS) Social Support Survey - Positive Social Interaction Subscale Score (Both Cohorts)
Description: The MOS Social Support Survey - Positive social interaction subscale is a 3 item subscale. Answers are on a 5 point scale with options "none of the time", "a little of the time", "some of the time", "most of the time", and "all of the time". Possible scores range from 3 to 15. Higher scores reflect higher feelings of positive social interaction (more perceived positive social interaction). The MOS Social Support Survey - Positive social interaction subscale is administered in both cohort 1 (Baseline, Mid-treatment, Post-treatment, up to 3 months) and cohort 2 (Baseline, Mid-treatment, Post-treatment, up to 6 months).
Time Frame: up to 6 months
Reporting Status: Not Posted

12. Other Pre Specified Outcome: Mean Change in Psychological Wellbeing Scale Short Form - Environmental Mastery Subscale Score (Both Cohorts)
Description: The Psychological Wellbeing Scale (Short Form) - Environmental Mastery Subscale is a 3 item scale. Answers are on a 6 point scale with options "strongly disagree", "moderately disagree", "slightly disagree", "slightly agree", "moderately agree", and "strongly agree". Possible scores range from 3 to 18. Higher scores reflect higher levels of environmental mastery. The MOS Social Support Survey - Environmental Mastery subscale is administered in both cohort 1 (Baseline, Mid-treatment, Post-treatment, up to 3 months) and cohort 2 (Baseline, Mid-treatment, Post-treatment, up to 6 months).
Time Frame: up to 6 months
Reporting Status: Not Posted

13. Other Pre Specified Outcome: Mean Change in Psychological Wellbeing Scale Short Form - Personal Growth Subscale Score (Both Cohorts)
Description: The Psychological Wellbeing Scale (Short Form) - Personal Growth subscale is a 3 item scale. Answers are on a 6 point scale with options "strongly disagree", "moderately disagree", "slightly disagree", "slightly agree", "moderately agree", and "strongly agree". Possible scores range from 3 to 18. Higher scores reflect higher levels of personal growth. The Psychological Wellbeing Scale - Personal Growth subscale is administered in both cohort 1 (Baseline, Mid-treatment, Post-treatment, up to 3 months) and cohort 2 (Baseline, Mid-treatment, Post-treatment, up to 6 months).
Time Frame: up to 6 months
Reporting Status: Not Posted

14. Other Pre Specified Outcome: Mean Change in Psychological Wellbeing Scale Short Form - Self-Acceptance Subscale Score (Both Cohorts)
Description: The Psychological Wellbeing Scale (Short Form) - Self-Acceptance subscale is a 3 item scale. Answers are on a 6 point scale with options "strongly disagree", "moderately disagree", "slightly disagree", "slightly agree", "moderately agree", and "strongly agree". Possible scores range from 3 to 18. Higher scores reflect higher feelings of self-acceptance. The Psychological Wellbeing Scale - Self-Acceptance subscale is administered in both cohort 1 (Baseline, Mid-treatment, Post-treatment, up to 3 months) and cohort 2 (Baseline, Mid-treatment, Post-treatment, up to 6 months).
Time Frame: up to 6 months
Reporting Status: Not Posted

15. Other Pre Specified Outcome: Mean Change in Psychological Wellbeing Scale Short Form - Autonomy Subscale Score (Both Cohorts)
Description: The Psychological Wellbeing Scale (Short Form) - Autonomy Subscale is a 3 item scale. Answers are on a 6 point scale with options "strongly disagree", "moderately disagree", "slightly disagree", "slightly agree", "moderately agree", and "strongly agree". Possible scores range from 3 to 18. Higher scores reflect higher levels of autonomy. The Psychological Wellbeing Scale - Autonomy subscale is administered in both cohort 1 (Baseline, Mid-treatment, Post-treatment, up to 3 months) and cohort 2 (Baseline, Mid-treatment, Post-treatment, up to 6 months).
Time Frame: up to 6 months
Reporting Status: Not Posted

16. Other Pre Specified Outcome: Mean Change in Psychological Wellbeing Scale Short Form - Purpose in Life Subscale Score (Both Cohorts)
Description: The Psychological Wellbeing Scale (Short Form) - Purpose in Life subscale is a 3 item scale. Answers are on a 6 point scale with options "strongly disagree", "moderately disagree", "slightly disagree", "slightly agree", "moderately agree", and "strongly agree". Possible scores range from 3 to 18. Higher scores reflect higher feelings of purpose in life. The Psychological Wellbeing Scale - Purpose in Life subscale is administered in both cohort 1 (Baseline, Mid-treatment, Post-treatment, up to 3 months) and cohort 2 (Baseline, Mid-treatment, Post-treatment, up to 6 months).
Time Frame: up to 6 months
Reporting Status: Not Posted

17. Other Pre Specified Outcome: Mean Change in Psychological Wellbeing Scale Short Form - Positive Relationships Subscale Score (Both Cohorts)
Description: The Psychological Wellbeing Scale (Short Form) - Positive Relationships subscale is a 3 item scale. Answers are on a 6 point scale with options "strongly disagree", "moderately disagree", "slightly disagree", "slightly agree", "moderately agree", and "strongly agree". Possible scores range from 3 to 18. Higher scores reflect higher levels of positive relationships. The Psychological Wellbeing Scale - Positive Relationships subscale is administered in both cohort 1 (Baseline, Mid-treatment, Post-treatment, up to 3 months) and cohort 2 (Baseline, Mid-treatment, Post-treatment, up to 6 months).
Time Frame: up to 6 months
Reporting Status: Not Posted

18. Other Pre Specified Outcome: Qualitative Summaries of Participant Experience in Post-Treatment Feedback (Both Cohorts)
Description: This qualitative data will be collected post-treatment from clients and clinicians. Focus groups and individual interviews will discuss usage of the platform and any feedback participants may have. Feedback from participants will be summarized to include common themes regarding likes and dislikes of the platform, implementation within the clinical setting, and participant ideas for future directions. Feedback is elicited at post-treatment in both cohort 1 (Month 3) and cohort 2 (Month 6).
Time Frame: up to 6 months
Reporting Status: Not Posted

19. Other Pre Specified Outcome: Quantitative Summaries of Participant Experience in Post-Treatment Feedback (Both Cohorts)
Description: This quantitative data will be collected post-treatment from clients and clinicians. Feedback forms will prompt participants to answer questions regarding their experience with the platform on a scale of 1 to 5, with higher scores reflecting a more positive experience. Frequency counts will be included here. Feedback is elicited at post-treatment in both cohort 1 (Month 3) and cohort 2 (Month 6).
Time Frame: up to 6 months
Reporting Status: Not Posted

20. Other Pre Specified Outcome: Mean Change in Questionnaire About the Process of Recovery - Total Score (Cohort 2 Only)
Description: The Questionnaire about the Process of Recovery (QPR) - Total Score is a 15-item scale. Answers are rated on a 5-point scale with options "disagree strongly", "disagree", "neither agree nor disagree", "agree", and "agree strongly. Possible scores range from 0 to 60. Higher scores are indicative of recovery. The QPR is administered in only cohort 2 (Baseline, Mid-treatment, Post-treatment, up to 6 months).
Time Frame: up to 6 months
Reporting Status: Not Posted

21. Other Pre Specified Outcome: Mean Change in Modified Colorado Symptom Index - Total Score (Cohort 2 Only)
Description: The Modified Colorado Symptom Index - Total Score is a 14-item scale. Answers are rated on a 4-point scale with options "not at all", "once during the month", "several times during the month", "several times a week", and "at least every day". Possible scores range from 0 to 56. Higher scores indicate greater emotional distress. The Modified Colorado Symptom Index is administered in only cohort 2 (Baseline, Mid-treatment, Post-treatment, up to 6 months).
Time Frame: up to 6 months
Reporting Status: Not Posted

22. Other Pre Specified Outcome: Mean Change in Social Anxiety Scale for Social Media Users - Total Score (Cohort 2 Only)
Description: The Social Anxiety Scale for Social Media Users (SAS-SMU) - Total Score is a 21-item scale. Answers are rated on a 5-point scale with options "never", "rarely", "sometimes", "often", and "always". Possible scores range from 21 to 105. Higher scores reflect greater anxiety related to social media usage. The SAS-SMU is administered in only cohort 2 (Baseline, Mid-treatment, Post-treatment, up to 6 months).
Time Frame: up to 6 months
Reporting Status: Not Posted

23. Other Pre Specified Outcome: Mean Change in Social Anxiety Scale for Social Media Users - Shared Content Anxiety Subscale Score (Cohort 2 Only)
Description: The Social Anxiety Scale for Social Media Users (SAS-SMU) - Shared Content Anxiety subscale is a 7-item scale. Answers are rated on a 5-point scale with options "never", "rarely", "sometimes", "often", and "always". Possible scores range from 7 to 35. Higher scores reflect greater anxiety related to sharing or creating content on social media. The SAS-SMU - Shared Content Anxiety subscale is administered in only cohort 2 (Baseline, Mid-treatment, Post-treatment, up to 6 months).
Time Frame: up to 6 months
Reporting Status: Not Posted

24. Other Pre Specified Outcome: Mean Change in Social Anxiety Scale for Social Media Users - Privacy Concern Anxiety Subscale Score (Cohort 2 Only)
Description: The Social Anxiety Scale for Social Media Users (SAS-SMU) - Privacy Concern Anxiety subscale is a 5-item scale. Answers are rated on a 5-point scale with options "never", "rarely", "sometimes", "often", and "always". Possible scores range from 5 to 25. Higher scores reflect greater anxiety related to privacy concerns on social media. The SAS-SMU - Privacy Concern Anxiety subscale is administered in only cohort 2 (Baseline, Mid-treatment, Post-treatment, up to 6 months).
Time Frame: up to 6 months
Reporting Status: Not Posted

25. Other Pre Specified Outcome: Mean Change in Social Anxiety Scale for Social Media Users - Interaction Anxiety Subscale Score (Cohort 2 Only)
Description: The Social Anxiety Scale for Social Media Users (SAS-SMU) - Interaction Anxiety subscale is a 6-item scale. Answers are rated on a 5-point scale with options "never", "rarely", "sometimes", "often", and "always". Possible scores range from 6 to 30. Higher scores reflect greater anxiety related to social interactions over social media. The SAS-SMU - Interaction Anxiety subscale is administered in only cohort 2 (Baseline, Mid-treatment, Post-treatment, up to 6 months).
Time Frame: up to 6 months
Reporting Status: Not Posted

26. Other Pre Specified Outcome: Mean Change in Social Anxiety Scale for Social Media Users - Self-Evaluation Anxiety Subscale Score (Cohort 2 Only)
Description: The Social Anxiety Scale for Social Media Users (SAS-SMU) - Self-Evaluation Anxiety subscale is a 3-item scale. Answers are rated on a 5-point scale with options "never", "rarely", "sometimes", "often", and "always". Possible scores range from 3 to 15. Higher scores reflect greater anxiety related to negative self-evaluation. The SAS-SMU - Self-Evaluation Anxiety subscale is administered in only cohort 2 (Baseline, Mid-treatment, Post-treatment, up to 6 months).
Time Frame: up to 6 months
Reporting Status: Not Posted

27. Other Pre Specified Outcome: Mean Change in Perceived Autonomy Support Scale - Total Score (Both Cohorts)
Description: The Perceived Autonomy Support Scale - Total Score is a 6-item scale. Answer are on a 7-point scale with options "strongly disagree", "moderately disagree", "slightly disagree", "neutral", "slightly agree", "moderately agree", and "strongly agree". Possible scores range from 6 to 42. Higher scores reflect greater perceived autonomy support. The Perceived Autonomy Support Scale is administered in both cohort 1 (Mid-treatment, Post-treatment, up to 6 weeks) and cohort 2 (1.5 Months, Mid-treatment, 4.5 Months, Post-treatment, up to 20 weeks).
Time Frame: up to 20 weeks
Reporting Status: Not Posted

28. Other Pre Specified Outcome: Mean Change in Twente Engagement With E-health Technologies Scale - Total Score (Cohort 2 Only)
Description: The Twente Engagement with E-health Technologies Scale - Total Score is a 9-item scale. Answers are on a 5-point scale with options "strongly disagree", "disagree", "neutral", "agree", and "strongly agree". Possible scores range from 0 to 36. Higher scores reflect greater engagement. The Twente Engagement with E-health Technologies Scale is administered in only cohort 2 (Baseline, 1.5 Months, Mid-treatment, 4.5 Months, Post-treatment, up to 6 months).
Time Frame: up to 6 months
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: From the time of signing informed consent through the end of post treatment, approximately 3 months for Cohort 1 and 6 months for Cohort 2.
Description: Since FEP Clinicians were not exposed to the study intervention, adverse events were not collected for this group.
Groups:
- FEP Clients (Cohort 2): Participants with first episode psychosis (FEP) recruited from First Episode Clinics in North Carolina (OASIS, Encompass, Eagle, and SHORE). Participants will use the online platform Horyzons for 6 months (cohort 2) as a part of their care plan. Participants will be encouraged to use both the therapeutic content and the moderated online community throughout their time in the study.
  Horyzons USA: Participants will be oriented to the site (online platform) and how to use it. The site includes curated therapeutic content surrounding issues such as generalized anxiety, social anxiety, social functioning, depression, and distress tolerance. The site also includes a social media function, in which participants and peer support specialists can post text, images, and videos. The site is monitored by graduate students and trained clinicians.
Arm/Group | FEP Clients (Cohort 1) | FEP Clients (Cohort 2)
All-Cause Mortality (participants affected / at risk) | 0/25 | 1/37
Serious Adverse Events (participants affected / at risk) | 1/25 | 0/37
Other Adverse Events (participants affected / at risk) | 0/25 | 0/37
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | FEP Clients (Cohort 1) (N=25) | FEP Clients (Cohort 2) (N=37)
Hospitalization for substance abuse (Psychiatric disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-10-26): https://cdn.clinicaltrials.gov/large-docs/51/NCT04673851/Prot_SAP_000.pdf